CLINICAL TRIAL: NCT01460342
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Parallel-Design, Study to Evaluate the Efficacy and Safety of Tadalafil Once-a-day Dosing for 12 Weeks in Asian Men With Signs and Symptoms of Benign Prostatic Hyperplasia
Brief Title: Phase 3 Study of Tadalafil Once-Daily in Asian Men With Benign Prostatic Hyperplasia (BPH)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14101; H6D-JE-LVJF (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-10-24; First posted 2011-10-26 (Estimated); Results first posted 2013-09-25 (Estimated); Last update posted 2013-09-25 (Estimated); Status verified 2013-07

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Prostatic hyperplasia; Benign prostatic hyperplasia; Lower urinary tract
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Following the 4-week placebo lead-in period, this arm will consist of a 12-week placebo treatment period involving 2 x 2.5-milligram (mg) tadalafil placebo tablets taken orally once daily.
  Interventions: Drug: Placebo
- Tadalafil (Experimental): Following the 4-week placebo lead-in period, this arm will consist of a 12-week treatment period involving 2 x 2.5-mg tadalafil tablets taken orally once daily.
  Interventions: Drug: Tadalafil; Drug: Placebo

INTERVENTIONS:
Drug: Tadalafil — 5 mg (2 x 2.5-mg tablets), given once daily as oral tablet
  Other Names: Cialis; LY450190
  Arms: Tadalafil
Drug: Placebo — 2 tablets (identical to 2.5-mg tadalafil tablets) given orally once daily.

SUMMARY:
This is a phase 3, randomized, double-blind, placebo-controlled, parallel-design, multinational study to evaluate the efficacy and safety of tadalafil once-a-day dosing for 12 weeks in Asian men with signs and symptoms of benign prostatic hyperplasia.

DETAILED DESCRIPTION:
Tadalafil is being investigated as a treatment for men with signs and symptoms of benign prostatic hyperplasia [BPH; also referred to as urinary disturbance or BPH-LUTS (BPH-lower urinary tract symptoms)] in Japan and overseas. Overseas studies and the Japanese dose-finding study LVIA (NCT00783094) identified tadalafil 5 mg once-daily as the recommended dose. The long-term safety and maintenance of effect was confirmed in the open-label extension of study LVIA. The risk-benefit profile was further studied in the Asian study LVHB (NCT00861757).

This study, LVJF, is to confirm the efficacy and safety of tadalafil 5 mg once-daily in Asian men with BPH-LUTS.

ELIGIBILITY:
Inclusion Criteria:

* Present with benign prostatic hyperplasia (BPH; also referred to as BPH-LUTS), based on the disease diagnostic criteria, at study entry.
* Provide signed informed consent at study entry.
* Have BPH-LUTS with a Total International Prostate Symptom Score (IPSS) of ≥13 at beginning of placebo lead-in period.
* Have bladder outlet obstruction of intermediate severity as defined by a urinary peak flow rate (Qmax) of ≥4 to ≤15 milliliters per second (mL/sec) [from a prevoid total bladder volume (assessed by ultrasound) of ≥150 to ≤550 milliliters (mL) and a minimum voided volume of 125 mL] at beginning of placebo lead-in period.
* Have prostate volume ≥20 mL estimated by transabdominal or transrectal ultrasound at study entry.
* Agree not to use any other approved or experimental pharmacologic BPH, erectile dysfunction (ED) and/or overactive bladder (OAB) treatments, including alpha-blockers, 5-alpha reductase inhibitors (5-ARIs), phosphodiesterase type 5 (PDE5) inhibitors, or herbal preparations at any time during the study.
* Have not taken the following treatments within the indicated duration:

  * Finasteride therapy for at least 3 months prior to beginning of placebo lead-in period.
  * Dutasteride therapy for at least 6 months prior to beginning of placebo lead-in period.
  * Anti-androgenic hormone therapy at least 12 months prior to beginning of placebo lead-in period.
  * All other BPH therapy (including herbal preparations) for at least 4 weeks prior to beginning of placebo lead-in period.
  * ED therapy for at least 4 weeks prior to beginning of placebo lead-in period.
  * OAB therapy for at least 4 weeks prior to beginning of placebo lead-in period.
* Demonstrate compliance with study drug administration requirements during the placebo lead-in period by administering ≥70% of prescribed doses, confirmed by documentation that the participant returned ≤30% of prescribed doses at randomization.

Exclusion Criteria:

* Prostate-specific antigen (PSA) >10.0 nanograms per milliliter (ng/mL) at study entry.
* PSA ≥4.0 to ≤10.0 ng/mL at study entry, if prostate malignancy has not been ruled out to the satisfaction of an urologist.
* Bladder postvoid residual (PVR) ≥300 mL by ultrasound determination at study entry.
* History of any of the following pelvic conditions (checked at study entry):

  * Pelvic surgery or any other pelvic procedure, including radical prostatectomy, pelvic surgery for removal of malignancy, or bowel resection.
  * Pelvic radiotherapy.
  * Any pelvic surgical procedure on the urinary tract, including minimally invasive BPH-LUTS therapies and penile implant surgery.
  * Lower urinary tract malignancy or trauma.
* Lower urinary tract instrumentation (including prostate biopsy) within 30 day of study entry.
* History of urinary retention or lower urinary tract (bladder) stones within 6 months of study entry.
* History of urethral obstruction due to stricture, valves, sclerosis, or tumor.
* Current neurologic disease or condition associated with neurogenic bladder (for example, Parkinson's disease, multiple sclerosis) at study entry.
* Clinical evidence of prostate cancer.
* Clinical evidence of any of the following bladder conditions:

  * Mullerian duct cysts.
  * Atonic, decompensated, or hypocontractile bladder.
  * Detrusor-sphincter dyssynergia (contraction of the detrusor without sphincter relaxation).
  * Intravesical obstruction (for example, intravesical median lobe of the prostate).
  * Interstitial cystitis.
* Clinical evidence of any of the following urinary tract conditions at study entry:

  * Urinary tract infection.
  * Urinary tract inflammation (including prostatitis). Urinary tract infection/inflammation is defined as a positive result for leukocyte esterase from a urine dipstick or >5 white blood cells (WBCs) per high-powered field on urinalysis from a centrifuged, clean-catch, midstream urine specimen.
  * Current antibiotic therapy for urinary tract infection.
  * Clinically significant microscopic hematuria as determined by an urologist.
* History of significant renal insufficiency, defined as receiving renal dialysis or having an estimated creatinine clearance <30 milliliters per minute (mL/min) at study entry, as calculated by the central laboratory using the Cockcroft-Gault formula.
* Clinical evidence of severe hepatic impairment [aspartate transaminase (AST) or alanine transaminase (ALT) >3-fold of the upper limit of normal range] at study entry.
* History of any of the following cardiac conditions (checked at study entry):

  * Angina requiring treatment with long-acting nitrates.
  * Angina requiring treatment with short-acting nitrates within 90 days of study entry.
  * Unstable angina within 90 days of study entry.
  * Positive cardiac stress test without documented evidence of subsequent, effective cardiac intervention.
* History of any of the following coronary conditions within 90 days of study entry:

  * Myocardial infarction.
  * Coronary artery bypass graft surgery.
  * Percutaneous coronary intervention (for example, angioplasty or stent placement).
* Any evidence of heart disease [New York Heart Association (NYHA) ≥Class III] within 6 months of study entry.
* Systolic blood pressure >160 or <90 millimeters of mercury (mm Hg) or diastolic blood pressure >100 or <50 mm Hg at study entry (if stress is suspected, retest under basal conditions), or malignant hypertension.
* Glycosylated hemoglobin (HbA1c) >9% at study entry.
* Scheduled or planned surgery (or any procedure requiring general, spinal, or epidural anesthesia) during the course of the study.
* History of significant central nervous system injuries (including stroke or spinal cord injury) within 6 months of study entry.
* History of drug, alcohol, or substance abuse within 6 months of study entry.
* Current treatment with nitrates, androgens, antiandrogens, estrogens, luteinizing hormone-releasing hormone agonists/antagonists, or anabolic steroids at study entry.
* Current systemic treatment with any of the following:

  * Potent cytochrome P450 3A4 (CYP3A4) inhibitors, such as ketoconazole or ritonavir.
  * CYP3A4 inducers such as rifampicin.
* Known or suspected to be hypersensitive to tadalafil, or any study drug components.
* Any conditions that would interfere with a participant's ability to provide informed consent or comply with study instructions, would place participant at increased risk, or might confound the interpretation of the study results.
* Previously completed or withdrawn from this study or any other study investigating tadalafil.
* Received treatment within the last 30 days with a drug or device that has not received regulatory approval for any indications at the time of informed consent. Participants who have been screen failures in previous studies may be eligible.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 610 (Actual)
Dates: Start 2011-12; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (17):
- Japan (11):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ehime
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyōgo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kagoshima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kyoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saitama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yamanashi
- South Korea (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Goyang-si
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Incheon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jeonju
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kwangju
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pusan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul

REFERENCES:
- [Derived] Takeda M, Yokoyama O, Lee SW, Murakami M, Morisaki Y, Viktrup L. Tadalafil 5 mg once-daily therapy for men with lower urinary tract symptoms suggestive of benign prostatic hyperplasia: results from a randomized, double-blind, placebo-controlled trial carried out in Japan and Korea. Int J Urol. 2014 Jul;21(7):670-5. doi: 10.1111/iju.12410. Epub 2014 Feb 27. PMID 24571205

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consisted of 3 periods: a screening/wash-out period (pre-randomization, 1 day up to 4 weeks), a placebo lead-in period (pre-randomization, 4 weeks, participant-blinded), and a double-blind treatment period (post-randomization, 12 weeks).
Groups:
- Placebo: Placebo: 2 tablets [identical to 2.5-milligram (mg) tadalafil tablets] given orally once daily for 4 weeks, during the placebo lead-in period and for 12 weeks, during the double-blind treatment period.
- Tadalafil: Tadalafil: 5 mg (two 2.5-mg tablets), given orally once daily for 12 weeks, during the double-blind treatment period. This followed a 4-week placebo lead-in period [2 tablets (identical to 2.5-mg tadalafil tablets) given orally once daily].
Period: Overall Study
Arm/Group | Placebo | Tadalafil
Started | 304 | 306
Received at Least 1 Dose of Study Drug | 304 | 306
Completed | 293 | 292
Not Completed | 11 | 14
Not completed — Adverse Event | 5 | 4
Not completed — Lost to Follow-up | 1 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Physician Decision | 1 | 3
Not completed — Lack of Efficacy | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tadalafil | Total
Number analyzed (Participants) | 304 | 306 | 610
Age Continuous [Mean (Standard Deviation); unit: years] | 60.9 (8.1) | 60.8 (7.7) | 60.9 (7.9)
Age, Customized [Number; unit: participants]
  <65 years | 201 | 198 | 399
  >=65 years | 103 | 108 | 211
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 304 | 306 | 610
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 304 | 306 | 610
Region of Enrollment [Number; unit: participants]
  Japan | 222 | 227 | 449
  Korea, Republic of | 82 | 79 | 161
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per square meter (kg/m^2)] — BMI was an estimate of body fat based on body weight divided by height squared.
  kilograms per square meter (kg/m^2) | 24.1 (2.9) | 24.0 (3.0) | 24.0 (3.0)
Current Tobacco Use [Number; unit: participants]
  Yes | 55 | 57 | 112
  No | 249 | 249 | 498
Alcohol Use [Number; unit: participants]
  Yes | 196 | 206 | 402
  No | 108 | 100 | 208
Benign Prostatic Hyperplasia (BPH) Severity [Number; unit: participants] — BPH severity rated mild [an International Prostate Symptom Score (IPSS) Total Score from 0 to 7], moderate (IPSS Total Score from 8 to 19), or severe (an IPSS Total Score >=20). The IPSS Total Score was the sum of Questions 1 through 7 in the IPSS questionnaire. Each question was based on the participant's urination experiences and prostate symptoms during the last month. Scores ranged from 0 (none/no symptoms) to 5 (frequent symptoms) for an IPSS Total Score that ranged from 0 to 35; higher numerical scores represented a greater severity of symptoms.
  participants
    Mild (IPSS Total Score 0 to 7) | 5 | 6 | 11
    Moderate (IPSS Total Score 8 to 19) | 167 | 166 | 333
    Severe (IPSS Total Score >=20) | 132 | 134 | 266
Duration of BPH [Mean (Standard Deviation); unit: years] | 4.0 (3.3) | 4.1 (3.2) | 4.0 (3.2)
Patient Global Impression of Severity (PGI-S) Scale [Number; unit: participants] — The PGI-S Scale measured the participant's perception of severity of illness at the time of assessment. Scores were 1 (Normal), 2 (Mild), 3 (Moderate), and 4 (Severe).
  participants
    Normal | 0 | 0 | 0
    Mild | 67 | 64 | 131
    Moderate | 187 | 195 | 382
    Severe | 50 | 47 | 97
Clinical Global Impression of Severity (CGI-S) Scale [Number; unit: participants] — The CGI-S Scale measured the clinician's perception of severity of illness at the time of the assessment. Scores were 1 (Normal), 2 (Mild), 3 (Moderate), and 4 (Severe).
  participants
    Normal | 0 | 0 | 0
    Mild | 33 | 41 | 74
    Moderate | 218 | 211 | 429
    Severe | 53 | 54 | 107
Previous Alpha-Blocker Therapy [Number; unit: participants] — Previous alpha-blocker therapy during the 12 months prior to study enrollment.
  participants
    Yes | 43 | 39 | 82
    No | 261 | 267 | 528
Previous Benign Prostatic Hyperplasia - Lower Urinary Tract Symptoms (BPH-LUTS) Therapy [Number; unit: Participants] — Previous BPH-LUTS therapy during the 12 months prior to study enrollment. Alpha-blocker therapy excluded.
  Participants
    Yes | 21 | 22 | 43
    No | 283 | 284 | 567
Postvoid Residual Volume (PVR) [Mean (Standard Deviation); unit: milliliters (mL)] — PVR was defined as the volume of urine remaining in the bladder after voiding, estimated by ultrasound.
  milliliters (mL) | 32.7 (50.0) | 26.9 (37.7) | 29.8 (44.3)
Prostate Volume [Mean (Standard Deviation); unit: mL] — The volume of prostate, estimated by transabdominal or transrectal ultrasound.
  mL | 31.6 (9.5) | 30.7 (8.5) | 31.1 (9.0)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Score of International Prostate Symptom Score (IPSS) at 12 Weeks
Description: The IPSS Total Score was the sum of Questions 1 through 7 in the IPSS questionnaire. Each question was based on the participant's urination experiences and prostate symptoms during the last month. Scores ranged from 0 (none/no symptoms) to 5 (frequent symptoms) for an IPSS Total Score that ranged from 0 to 35; higher numerical scores represented a greater severity of symptoms. Least squares (LS) mean was based on the mixed-effect model repeated measures (MMRM) model analysis with participants as random effects, treatment, prior alpha-blocker use (yes/no), country (Japan/Korea), visit, and treatment-by-visit interaction as fixed effects, and baseline value and placebo lead-in total IPSS change as fixed covariates.
Time Frame: Baseline, 12 weeks
Population: Randomized participants who received at least 1 dose of study drug and had non-missing data at baseline.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 301 | 305
units on a scale | -4.5 (0.4) | -6.0 (0.4)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -1.5, 95% CI 2-sided [-2.4 to -0.6], Standard Error of Mean 0.5

2. Secondary Outcome: Change From Baseline in Total Score of International Prostate Symptom Score (IPSS)
Description: as for outcome 1
Time Frame: Baseline, 4 weeks, 8 weeks
Population: Randomized participants who received at least 1 dose of study drug and had non-missing data at baseline.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 301 | 305
units on a scale
  Change at Week 4 | -2.8 (0.3) | -4.0 (0.4)
  Change at Week 8 | -4.0 (0.4) | -5.2 (0.4)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The p-value is for the change from baseline in the IPSS Total Score at Week 4; Mean Difference (Final Values) = -1.3, 95% CI 2-sided [-2.0 to -0.5], Standard Error of Mean 0.4
Statistical Analysis 2: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis — The p-value is for the change from baseline in the IPSS Total Score at Week 8; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-2.0 to -0.4], Standard Error of Mean 0.4

3. Secondary Outcome: Change From Baseline in the International Prostate Symptom Score (IPSS) Storage (Irritative) Subscore
Description: The IPSS Storage (Irritative) Subscore was the sum of Questions 2, 4, and 7 in the IPSS questionnaire. Each question was scored from 0 (no irritative symptoms) to 5 (frequent irritative symptoms) for an IPSS Storage (Irritative) Subscore that ranged from 0 to 15; higher numerical scores represented a greater severity of symptoms. Least squares (LS) mean was based on the mixed-effect model repeated measures (MMRM) model analysis with participants as random effects, treatment, prior alpha-blocker use (yes/no), country (Japan/Korea), visit, and treatment-by-visit interaction as fixed effects, and baseline value and placebo lead-in total IPSS change as fixed covariates.
Time Frame: Baseline, 4 weeks, 8 weeks, 12 weeks
Population: Randomized participants who received at least 1 dose of study drug and had non-missing data at baseline.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 301 | 305
units on a scale
  Change at 4 Weeks | -0.9 (0.1) | -1.2 (0.2)
  Change at 8 Weeks | -1.3 (0.2) | -1.7 (0.2)
  Change at 12 Weeks | -1.4 (0.2) | -2.0 (0.2)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.090, Mixed Models Analysis — The p-value was for the change from baseline in the IPSS Storage (Irritative) Subscore at Week 4; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.6 to 0.0], Standard Error of Mean 0.2
Statistical Analysis 2: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.011, Mixed Models Analysis — The p-value was for the change from baseline in the IPSS Storage (Irritative) Subscore at Week 8; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-0.8 to -0.1], Standard Error of Mean 0.2
Statistical Analysis 3: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis — The p-value was for the change from baseline in the IPSS Storage (Irritative) Subscore at Week 12; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-0.9 to -0.2], Standard Error of Mean 0.2

4. Secondary Outcome: Change From Baseline in the International Prostate Symptom Score (IPSS) Voiding (Obstructive) Subscore
Description: The IPSS Voiding (Obstructive) Subscore was the sum of Questions 1, 3, 5, and 6 in the IPSS questionnaire. Each question was scored from 0 (no obstructive symptoms) to 5 (frequent obstructive symptoms) for an IPSS Voiding (Obstructive) Subscore that ranged from 0 to 20; higher numerical scores represented a greater severity of symptoms. Least squares (LS) mean was based on the mixed-effect model repeated measures (MMRM) model analysis with participants as random effects, treatment, prior alpha-blocker use (yes/no), country (Japan/Korea), visit, and treatment-by-visit interaction as fixed effects, and baseline value and placebo lead-in total IPSS change as fixed covariates.
Time Frame: Baseline, 4 weeks, 8 weeks, 12 weeks
Population: Randomized participants who received at least 1 dose of study drug and had non-missing data at baseline.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 301 | 305
units on a scale
  Change at Week 4 | -1.8 (0.2) | -2.8 (0.2)
  Change at Week 8 | -2.6 (0.3) | -3.4 (0.3)
  Change at Week 12 | -3.1 (0.3) | -4.0 (0.3)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The p-value was for the change from baseline in the IPSS Voiding (Obstructive) Subscore at Week 4; Mean Difference (Final Values) = -1.0, 95% CI 2-sided [-1.5 to -0.4], Standard Error of Mean 0.3
Statistical Analysis 2: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.007, Mixed Models Analysis — The p-value was for the change from baseline in the IPSS Voiding (Obstructive) Subscore at Week 8; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-1.3 to -0.2], Standard Error of Mean 0.3
Statistical Analysis 3: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis — The p-value was for the change from baseline in the IPSS Voiding (Obstructive) Subscore at Week 12; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-1.5 to -0.3], Standard Error of Mean 0.3

5. Secondary Outcome: Change From Baseline in the International Prostate Symptom Score (IPSS) Quality of Life (QoL) Index
Description: The IPSS QoL Index assessed the participant's response to the following question, "If you were to spend the rest of your life with your urinary condition just the way it is now, how would you feel about that?". Response options were 0 (Delighted), 1 (Pleased), 2 (Mostly satisfied), 3 (Mixed, about equally satisfied and dissatisfied), 4 (Mostly dissatisfied), 5 (Unhappy), and 6 (Terrible), for a QoL Index Score that ranged from 0 to 6. Least squares (LS) mean was based on the mixed-effect model repeated measures (MMRM) model analysis with participants as random effects, treatment, prior alpha-blocker use (yes/no), country (Japan/Korea), visit, and treatment-by-visit interaction as fixed effects, and baseline value and placebo lead-in total IPSS change as fixed covariates.
Time Frame: Baseline, 4 weeks, 8 weeks, 12 weeks
Population: Randomized participants who received at least 1 dose of study drug and had non-missing data at baseline.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 301 | 305
units on a scale
  Change at Week 4 | -0.5 (0.1) | -0.6 (0.1)
  Change at Week 8 | -0.7 (0.1) | -0.8 (0.1)
  Change at Week 12 | -0.9 (0.1) | -1.1 (0.1)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.277, Mixed Models Analysis — The p-value was for the change from baseline in the IPSS QoL Index Score at Week 4; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.2 to 0.1], Standard Error of Mean 0.1
Statistical Analysis 2: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.170, Mixed Models Analysis — The p-value was for the change from baseline in the IPSS QoL Index Score at Week 8; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.3 to 0.1], Standard Error of Mean 0.1
Statistical Analysis 3: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.038, Mixed Models Analysis — The p-value was for the change from baseline in the IPSS QoL Index Score at Week 12; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.4 to -0.0], Standard Error of Mean 0.1

6. Secondary Outcome: Patient Global Impression of Improvement (PGI-I) Scale at 12 Weeks
Description: The PGI-I scale measured the participant's perception of improvement at the time of assessment compared with the start of treatment. Scores were 1 (Very much better), 2 (Much improved), 3 (Minimally improved), 4 (No change), 5 (Minimally worse), 6 (Much worse), and 7 (Very much worse).
Time Frame: 12 Weeks
Population: Randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 304 | 306
participants
  Very Much Better | 9 | 18
  Much Better | 55 | 79
  A Little Better | 138 | 148
  No Change | 90 | 55
  A Little Worse | 7 | 2
  Much Worse | 0 | 0
  Very Much Worse | 2 | 0
  Missing | 3 | 4
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — The p-value was from the Cochran-Mantel-Haenszel test adjusted for baseline severity of benign prostatic hyperplasia lower urinary tract symptoms (BPH-LUTS) and previous alpha-blocker therapy

7. Secondary Outcome: Clinician Global Impression of Improvement (CGI-I) Scale at 12 Weeks
Description: The CGI-I measured the clinician's perception of participant improvement at the time of assessment compared with the start of treatment. Scores were 1 (Very much better), 2 (Much improved), 3 (Minimally improved), 4 (No change), 5 (Minimally worse), 6 (Much worse), and 7 (Very much worse).
Time Frame: 12 Weeks
Population: Randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 304 | 306
participants
  Very Much Improved | 10 | 14
  Much Improved | 74 | 103
  Minimally Improved | 115 | 125
  No Change | 93 | 59
  Minimally Worse | 8 | 1
  Much Worse | 0 | 0
  Very Much Worse | 1 | 0
  Missing | 3 | 4
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 6, analysis 1]

8. Secondary Outcome: Change From Baseline in Modified International Prostate Symptom Score (mIPSS) Score at 2 Weeks
Description: The mIPSS Total Score was the sum of Questions 1 through 7 in the mIPSS questionnaire, which was a modified version of the IPSS questionnaire. Questions about the participant's urination experiences and prostate symptoms in the IPSS questionnaire were modified to obtain responses based on time since the last visit rather than during the last month. Each question was scored from 0 (none/no symptoms) to 5 (frequent symptoms) for an mIPSS Total Score that ranged from 0 to 35; higher numerical scores represented a greater severity of symptoms. Least squares (LS) mean was based on the analysis of covariance (ANCOVA) model with treatment, prior alpha-blocker use (yes/no), and country (Japan/Korea) as fixed effects, and baseline value and placebo lead-in total IPSS change as fixed covariates.
Time Frame: Baseline, 2 weeks
Population: Randomized participants who received at least 1 dose of study drug and had non-missing data at baseline.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 301 | 305
units on a scale | -2.1 (0.3) | -2.7 (0.3)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.060, ANCOVA; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-1.2 to 0.0], Standard Error of Mean 0.3

ADVERSE EVENTS:
Arm/Group | Placebo | Tadalafil
Serious Adverse Events (participants affected / at risk) | 1/304 | 2/306
Other Adverse Events (participants affected / at risk) | 75/304 | 87/306
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=304) | Tadalafil (N=306)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0) — Event resulted in death within 30 days of study drug discontinuation
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=304) | Tadalafil (N=306)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Ear discomfort (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Asthenopia (Eye disorders) | 0 (0) | 1 (1)
Astigmatism (Eye disorders) | 0 (0) | 1 (1)
Erythema of eyelid (Eye disorders) | 0 (0) | 1 (1)
Eyelid oedema (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Vitreous detachment (Eye disorders) | 0 (0) | 1 (1)
Vitreous floaters (Eye disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 2 (3)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 5 (5)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 12 (12)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastritis atrophic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingivitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lip dry (Gastrointestinal disorders) | 1 (1) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 2 (2) | 0 (0)
Periodontitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Granuloma (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Therapeutic response unexpected (General disorders) | 0 (0) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 3 (3) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 10 (11) | 13 (14)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 3 (3)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Tracheitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (4) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 6 (6) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Blood chloride decreased (Investigations) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 7 (7) | 7 (7)
Blood sodium decreased (Investigations) | 0 (0) | 1 (1)
Blood urine (Investigations) | 1 (1) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 1 (1) | 4 (4)
Gamma-glutamyltransferase increased (Investigations) | 3 (3) | 1 (1)
Glucose urine present (Investigations) | 0 (0) | 2 (2)
White blood cell count decreased (Investigations) | 2 (2) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Burning sensation (Nervous system disorders) | 0 (0) | 1 (1)
Carotid arteriosclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 6 (6) | 9 (9)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Erection increased (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Spontaneous penile erection (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Electrocauterisation (Surgical and medical procedures) | 1 (1) | 0 (0)
Rectal polypectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 2 (2) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days